CLINICAL TRIAL: NCT06607614
Title: Prioritizing Resumption of Colorectal Screening After COVID
Brief Title: A Predictive Model Based on Quantitative Fecal Immunochemical Test Can Stratify the Risk of CRC in an Organized Screening Program
Acronym: PRIORITIZE
Status: Not yet recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: European Society of Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Silvia Pecere, M.D. PhD, Catholic University of the Sacred Heart
Other Study IDs: 6404
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Screening
Keywords: fecal immunochemical test; Colorectal cancer; screening program
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective cohort: All FIT+ patients of participating centers that are active in the CRC regional screening programs, with follow up colonscopies scheduled according to the developed scoring system.
  Interventions: Other: Colorectal Cancer Screening Fecal Immunochemical Test

INTERVENTIONS:
Other: Colorectal Cancer Screening Fecal Immunochemical Test — Fecal Immunochemical Test
  Other Names: Fecal Immunochemical Test

SUMMARY:
The COVID-19 pandemic has disrupted every aspect of medical care, including screening programs and preventive medical care . Organized FIT-based colorectal cancer screening programs make no exception, since their efficacy depends on a multi-tiered series of interventions that were hampered by the pandemic at multiple levels. In detail, the first level of intervention, namely population based FIT tests distributed to the population, has seen a dramatic decrease of number of tests performed for both organizational reasons (i.e. less personnel deployed to testing sites) and for failure to present fecal samples from patients for fear of contagion or impossibility to reach the drop-off sites for state-imposed limitations. Secondly, the referral of FIT positive patients to subsequent colonoscopy was stopped or delayed since endoscopy services have been undergoing only emergent and urgent procedures. Thirdly, patients diagnosed with advanced neoplasia or cancer have seen their endoscopic or surgical removal procedures delayed or canceled . Regarding post-FIT colonoscopy workup, European Screening Guidelines recommend a 30-day maximum span between a positive FIT test and subsequent colonoscopy. It is well known that any delay in post-FIT+ colonoscopy results in an increase in advanced neoplasia and colorectal cancer, that reaches dramatic levels after 6 months .

Our purpose is to develop and validate, using the quantitative level of faecal hemoglobin found in FIT, a simple scoring system to effectively sub-stratify CRC risk of FIT positive patients.

ELIGIBILITY:
Inclusion Criteria:

* All FIT+ patients awaiting to be scheduled for colonoscopy workup. Patients will be invited to undergo a colonoscopy, and depending on its outcome, patients are referred for surgery, postcolonoscopy surveillance, or further rounds of FIT.

Exclusion Criteria:

* Individuals with a prevalent diagnosis of CRC are excluded from the program, as well as patients that have already undergone a high quality colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FIT+, scheduled for colonoscopy
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer rate in the different risk groups | 12 months
  Colorectal cancer rate in the different risk groups

SECONDARY OUTCOMES:
Advanced adenoma rate in the different risk group | 12 months
  Advanced adenoma rate in the different risk group
Any adenoma rate in the different risk groups | 12 months
  Any adenoma rate in the different risk groups

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cubiella J, Digby J, Rodriguez-Alonso L, Vega P, Salve M, Diaz-Ondina M, Strachan JA, Mowat C, McDonald PJ, Carey FA, Godber IM, Younes HB, Rodriguez-Moranta F, Quintero E, Alvarez-Sanchez V, Fernandez-Banares F, Boadas J, Campo R, Bujanda L, Garayoa A, Ferrandez A, Pinol V, Rodriguez-Alcalde D, Guardiola J, Steele RJ, Fraser CG; COLONPREDICT study investigators. The fecal hemoglobin concentration, age and sex test score: Development and external validation of a simple prediction tool for colorectal cancer detection in symptomatic patients. Int J Cancer. 2017 May 15;140(10):2201-2211. doi: 10.1002/ijc.30639. Epub 2017 Mar 6. PMID 28187494
- [Background] Park CH, Jung YS, Kim NH, Park JH, Park DI, Sohn CI. Usefulness of risk stratification models for colorectal cancer based on fecal hemoglobin concentration and clinical risk factors. Gastrointest Endosc. 2019 Jun;89(6):1204-1211.e1. doi: 10.1016/j.gie.2019.02.023. Epub 2019 Feb 25. PMID 30817918
- [Background] Kim NH, Lim JW, Kim S, Lim JY, Kim W, Park JH, Park DI, Sohn CI, Jung YS. Association of time to colonoscopy after a positive fecal test result and fecal hemoglobin concentration with risk of advanced colorectal neoplasia. Dig Liver Dis. 2019 Apr;51(4):589-594. doi: 10.1016/j.dld.2018.12.008. Epub 2018 Dec 23. PMID 30733186
- [Background] Zorzi M, Hassan C, Capodaglio G, Baracco M, Antonelli G, Bovo E, Rugge M. Colonoscopy later than 270 days in a fecal immunochemical test-based population screening program is associated with higher prevalence of colorectal cancer. Endoscopy. 2020 Oct;52(10):871-876. doi: 10.1055/a-1159-0644. Epub 2020 Apr 30. PMID 32356282